CLINICAL TRIAL: NCT03712982
Title: Attention to Variability During Infertility
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Harvard University (Other)
Responsible Party: Principal Investigator, Karyn Gunnet-Shoval, Principal Investigator, Harvard University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Other
Other Study IDs: IRB16-1683
Record Dates: First submitted 2018-09-25; First posted 2018-10-19 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Infertility; Infertility, Female; Infertility, Male
Keywords: Infertility; Fertility; Mindfulness; Ellen Langer; Wellbeing; Attention to Variability
MeSH Terms: conditions — Infertility; Infertility, Female; Infertility, Male

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Waitlist Control (No Intervention): All participants in this condition will complete all measures online at three different points in time, including one narrative response at T2.
- Attention to Variability - Patient Only (Experimental): All participants in this condition will complete all measures online at three different points in time, including one narrative response at T2. They will also be instructed to complete a mindfulness intervention at home and respond to diary-type text messaging questions twice daily for two weeks (14 days).
  Interventions: Behavioral: Attention to Variability - Patient Only
- Attention to Variability - Partner Only (Experimental): All participants in this condition will complete all measures online at three different points in time, including one narrative response at T2. Partners of the infertile women will also be instructed to complete a mindfulness intervention at home and respond to diary-type text messaging questions twice daily for two weeks (14 days).
  Interventions: Behavioral: Attention to Variability - Partner Only
- Attention to Variability - Patient & Partner (Experimental): All participants in this condition will complete all measures online at three different points in time, including one narrative response at T2. All participants (patients and partners) will also be instructed to complete a mindfulness intervention at home and respond to diary-type text messaging questions twice daily for two weeks (14 days).
  Interventions: Behavioral: Attention to Variability - Patient & Partner
- Infertility Stories - Reading (Active Comparator): All participants in this condition will complete all measures online at three different points in time, including one narrative response at T2. They will also be instructed to do an at-home reading activity several times over a period of 2 weeks.
  Interventions: Other: Infertility Stories - Reading

INTERVENTIONS:
Behavioral: Attention to Variability - Patient Only — In Attention to Variability we ask the participant to attend to the natural fluctuations in mood and physiology that occur throughout the day, to notice when a symptom is better or worse and to ask why it may be.
  Arms: Attention to Variability - Patient Only
Behavioral: Attention to Variability - Partner Only — In Attention to Variability we ask the participant to attend to the natural fluctuations in mood and physiology in their partner that occur throughout the day, to notice when a symptom is better or worse and to ask why it may be.
  Arms: Attention to Variability - Partner Only
Behavioral: Attention to Variability - Patient & Partner — Same as patient and partner only conditions, just that in this condition both the patient and partner do their corresponding intervention rather than only one of them.
  Arms: Attention to Variability - Patient & Partner
Other: Infertility Stories - Reading — Reading Stories About Others' Infertility Experiences
  Other Names: Reading Activity
  Arms: Infertility Stories - Reading

SUMMARY:
Infertility affects approximately one in seven couples, and it can be a devastating diagnosis and difficult experience for couples to endure. Ellen Langer, Ph.D., Director of the Langer Lab at Harvard, has spent several decades demonstrating evidence supporting a mind-body approach to improve wellbeing and overall functioning. Specifically, she asserts that Mindfulness in its most basic sense - paying attention in the moment - is enough to create both perceived (e.g., self-reported) and real (e.g., objective testing) change. Langer and her colleague, for example, demonstrated that "Trait mindfulness predicted the well-being of expecting mothers and better neonatal outcomes. Mindfulness training resulted in better health for the expecting mother". In this study, Mindfulness training refers to "attention to sensation variability." Such interventions are cost effective, minimally invasive, less time-consuming for practitioners and participants and generally easy to learn.

Langer and her colleague's study refers to pregnancy. Infertility is unlike pregnancy in its exact clinical diagnosis. Nevertheless, similar to pregnancy, infertility is considered a clinical condition affecting the body, in this case the reproductive system. Therefore, based on the results of studies like Langer and her colleague's, that used participants with clinical conditions affecting the reproductive system, the investigators propose similar mindfulness intervention (attention to sensation variability) research with infertile individuals. However, the investigators intend to extend our examination to also include a treatment group with the partners of the infertile individuals, as little, if any research, has attempted to do so previously. The investigators hypothesize that state mindfulness (groups exposed to mindfulness intervention) will improve wellbeing in the infertile patient and her partner and that trait mindfulness will predict ability to become pregnant.

DETAILED DESCRIPTION:
Couples who have been trying to conceive for at least a year, have attended at least one doctor's appointment with an infertility/fertility specialist and have been advised by their physician to undergo their first IVF cycle will be recruited for this study.

Participants (couples) will be randomly assigned (assignment determined immediately following recruitment by a member of our research team), if eligible to one of four of five experimental conditions, which are described below. Assignment will occur on a 1:2:2:2:1 basis, such that for every two couples assigned to Conditions 2, 3 and 4 (mindfulness conditions) one couple will be assigned to Conditions 1 and 5 (control conditions). Couples will be told that we are interested in exploring if practicing mindful attention during the IVF process may improve patient and partner wellbeing during and following their first IVF cycle. All participants will be instructed to complete study measures, at three different points in time, via an online link.

ELIGIBILITY:
Inclusion criteria (infertile patients and their partners):

* 18+ years of age;
* Female patients who have been trying to conceive for at least a year, have attended at least one doctor's appointment with an infertility/fertility specialist and have been advised by their physician to undergo their first IVF cycle;
* Participants (patients and partners) with no known biological children.

Exclusion criteria (infertile patients and their partners):

* Individuals who do not meet the inclusion criteria above;
* Participants (patients and partners) with secondary infertility (already have a child);
* Participants (patients and partners) with a cut point score of less than 60 on the Mental Health Inventory (MHI-5) (assessed at phone screening).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2016-12-05 (Actual); Primary Completion 2022-12-05 (Estimated); Study Completion 2022-12-05 (Estimated)

PRIMARY OUTCOMES:
Patient and Partner Wellbeing - Langer Mindfulness Scale (LMS) | Approximately 8 minutes
  4 subscales, each ranging from 1-7, with 1 being 'Strongly Disagree' and 7 being 'Strongly Agree'. Subscales are 'Flexibility' (includes 4 items); 'Novelty Seeking' (6 items); 'Novelty Producing' (6 items); 'Engagement' (5 items). 7 items are reverse scored. To determine overall Mindfulness score, sum all items (items 1-21).
Patient and Partner Wellbeing - Positive and Negative Affect Schedule (PANAS) | Approximately 8 minutes
  Scale consists of a number of words that describe different feelings and emotions. Participants indicate to what extent they have a particular way in the past few hours. The scale ranges from 1 (Very slightly or not at all) to 5 (extremely).
  Individuals decide which of the 20 questions are positive and which are negative. Scores are then added for the 10 positive words and separately for the 10 negative words. The scores generated will vary along the scale of 10 - 50, with lower scores indicating low (positive or negative) affect and higher scores indicating high (positive or negative) affect.
Patient and Partner Wellbeing - Rosenberg Self-Esteem Scale (RSE) | Approximately 5 minutes
  A 10-item scale that measures global self-worth by measuring both positive and negative feelings about the self. The scale is believed to be unidimensional. All items are answered using a 4-point Likert scale format ranging from 1 (strongly agree) to 4 (strongly disagree).
  Scoring: Items 2, 5, 6, 8, 9 are reverse scored. Scores are then summed for all ten items on a continuous scale. Higher scores indicate higher self-esteem.
Patient and Partner Wellbeing - Satisfaction With Life Scale (SWLS) | Approximately 3 minutes
  A 5-item scale designed to measure global cognitive judgments of one's life satisfaction. Participants indicate how much they agree or disagree with each of the 5 items using a 7-point scale that ranges from 1 (strongly disagree) to 1 (strongly agree).
  Scoring : Scoring should be kept continuous (scores are summed up on each item).
Patient and Partner Wellbeing - Perceived Stress Scale (PSS) | Approximately 5 minutes
  The following questions ask about one's feelings and thoughts during the past month. In each question, individuals are asked how often they felt or thought a certain way.
  Scoring: Each item is rated on a 5-point scale ranging from (0) never to (4) almost always. Positively worded items are reverse scored, and the ratings are summed, with higher scores indicating more perceived stress. PSS-10 scores are obtained by reversing the scores on the four positive items: For example, 0=4, 1=3, 2=2, etc. and then summing across all 10 items. Items 4, 5, 7, and 8 are the positively stated items.
Patient and Partner Wellbeing - Couples Satisfaction Index (CSI) | Approximately 11 minutes
  A 32-item scale designed to measure one's satisfaction in a relationship. The scale has a variety of items with different response scales and formats.
  Question Scoring:
  1: 0 (Extremely Unhappy) to 6 (Perfect); 2-4: 0 (Always Disagree) to 5 (Always Agree); 5: 0 (Never) to 5 (All the time); 6: 0 (All the time) to 5 (Never); 7-18: 0 (Not at all True) to 5 (Completely True); 19-22: 0 (Not at All) to 5 (Completely); 23: 0 (Worse than all others [extremely bad]) to 5 (Better than all others [extremely good]); 24-25: 0 (Never) - 5 (More Often); 26: 0 (Boring) to 5 (Interesting); 27: 0 (Bad) to 5 (Good); 28: 0 (Empty) to 5 (Full); 29: 0 (Lonely) to 5 (Friendly); 30: 0 (Fragile) to Sturdy (5); 31: 0 (Discouraging) to 5 (Hopeful); 32: 0 (Miserable) to 5 (Enjoyable).
Patient and Partner Wellbeing - Tolerance of Ambiguity Scale | Approximately 10 minutes
  The instrument consists of 16 items on a scale ranging from 1 (Strongly Disagree) to 7 (Strongly Agree).
  High scores indicate a greater intolerance for ambiguity. To score the instrument, the even-numbered items must be reverse-scored. Three subscales can also be computed to reveal the major source of intolerance of ambiguity - novelty (N), complexity (c), or insolubility (I).
  Having intolerance of ambiguity means that an individual tends to perceive situations as threatening rather than promising. Lack of information or uncertainty, for example, would make such a person uncomfortable. Ambiguity arises from three main sources: novelty, complexity and insolubility.
Patient and Partner Wellbeing - Narrative question about their mind-body experience | Approximately 8 minutes
  Narrative question about their mind-body experience over the past three weeks

SECONDARY OUTCOMES:
Ability to become pregnant | 2 minutes
  Question about whether or not they got pregnant

CONTACTS AND LOCATIONS:
Overall Officials: Karyn Gunnet-Shoval, PhD, Principal Investigator — Harvard University; Katherine Bercovitz, Principal Investigator — Harvard University; Ellen Langer, PhD, Study Director — Harvard University
Locations (1):
- Boston IVF/IVF New England, Waltham, Massachusetts, United States

REFERENCES:
- [Result] Zilcha-Mano S, Langer E. Mindful Attention to Variability Intervention and Successful Pregnancy Outcomes. J Clin Psychol. 2016 Sep;72(9):897-907. doi: 10.1002/jclp.22294. Epub 2016 Mar 23. PMID 27007939